CLINICAL TRIAL: NCT02296840
Title: Comparing Narcotics With Non-steroidal Anti-inflammatory Drugs (NSAIDS) Post-operatively in Pediatric Patients Undergoing Adenotonsillectomy
Brief Title: Post-operative Pain Control After Pediatric Adenotonsillectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Roy Rajan, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00070851
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Tonsillitis; Obstructive Sleep Apnea; Sleep Disordered Breathing; Adverse Reaction to Drug
Keywords: analgesia; non-steroidal anti-inflammatory drugs; narcotic-containing pain medication
MeSH Terms: conditions — Tonsillitis; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Drug-Related Side Effects and Adverse Reactions; Agnosia | interventions — Ibuprofen; oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Experimental): After undergoing adenotonsillectomy, patients who are randomized into the test intervention arm will receive ibuprofen (10mg/kg/day every 6-8 hours) after surgery.
  Interventions: Drug: Ibuprofen
- Hydrocodone-acetaminophen (Control) (Active Comparator): After undergoing adenotonsillectomy, patients who are randomized into the control intervention will receive hydrocodone-acetaminophen (0.15mg/kg/day every 4-6 hours).
  Interventions: Drug: Hydrocodone-Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 10mg/kg/day every 6-8 hours
  Other Names: Advil; Motrin
  Arms: Ibuprofen
Drug: Hydrocodone-Acetaminophen — Hydrocodone-Acetaminophen 0.15mg/kg/day every 4-6 hours
  Other Names: Vicodin; Lortab
  Arms: Hydrocodone-acetaminophen (Control)

SUMMARY:
Adenotonsillectomy is one of the most common surgical procedures performed in the pediatric population in the United States. It is generally a well-tolerated procedure with post-operative bleeding risk ranging from 3-5% in children. Post-operative pain following adenotonsillectomy has significant morbidity and may result in prolonged hospital stay or re-admission to the hospital. Post-operative analgesia is most commonly managed with narcotic-containing pain medication. In recent years however, there is evidence that some patients may manifest increased sensitivity to narcotics, resulting in life-threatening respiratory compromise. Though there is a theoretical risk that nonsteroidal anti-inflammatory drugs (NSAIDs) increase bleeding time by disrupting platelet aggregation, evidence of detrimental effects (i.e. increased risk of postoperative bleeding) remains inconclusive for these generally well-tolerated medications. The goal of this study is to determine the incidence of post-operative bleeding and to determine the efficacy of NSAIDs in the management of post-operative pain following pediatric adenotonsillectomy, versus more commonly used narcotic pain medication. The study design will be an initial retrospective study to collect pilot data on the incidence of postoperative hemorrhage and indicators of adequate/inadequate pain control in children age 4 to 17 undergoing adenotonsillectomy. This will be followed by a prospective, randomized, single-blind controlled study in which orally-administered ibuprofen (test intervention) is compared to acetaminophen-hydrocodone (control intervention) in the postoperative period following adenotonsillectomy.

DETAILED DESCRIPTION:
Post-operative pain management in pediatric patients undergoing adenotonsillectomy is challenging not only for the child, but also for the clinician and caregiver. Uncontrolled pain carries a high level of morbidity and can result in prolonged hospital stay and/or readmission, dehydration, weight loss, and other undesirable effects. In light of recent high-profile controversies regarding the safety of codeine the search for effective and safe analgesia continues. The American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS) guidelines suggest that NSAIDs are safe to use in the post-operative period. Here, the investigators compare bleeding risk and pain control using acetominophen-hydrocodone (control) versus ibuprofen (intervention) in the post-operative period in pediatric patients undergoing adenotonsillectomy. The investigators hypothesize that ibuprofen will not be associated with increased bleeding risk and will control post-operative pain as well as acetominophen-hydrocodone.

Initial retrospective chart review (Data to be extracted from the patients' charts):

* Demographic data
* Surgical data
* Postoperative data
* Descriptive analysis to determine incidence of postoperative bleeding following adenotonsillectomy and its relation to demographic factors or surgical factors, incidence of postoperative pain problems and relation to demographic or surgical factors.

Prospective, randomized, single-blind trial:

* Study Group Allocation/Randomization: Study participants will be randomized into two post-operative pain medication treatment arms, using block randomization. Patients who are randomized into the test intervention arm will receive ibuprofen (10mg/kg/day every 6-8 hours) after surgery. Patients who are randomized into the control intervention will receive hydrocodone-acetaminophen (0.15mg/kg/day every 4-6 hours). This randomization will be performed by Ansley Roche MD, a co-investigator. The operating surgeons will be unaware of the group assignments at the time of randomization, at the time of surgery, and in the post-operative period. (The participant and caregiver will not be blinded to the type of post-operative pain medication they will receive.) Once a study participant has been randomized to group, the group assignment information will be provided to the otolaryngology resident at Egleston. The resident will write the appropriate prescription and provide this to the patient's family prior to discharge.
* Postoperative pain assessment: Using the Faces Pain Scale , the pediatric patient will indicate his/her pain level at scheduled intervals. Pain level will be recorded by the caregiver and pain medication will be administered appropriately based on level of patient's self-reported pain. A log of pain medication administered will be kept for each dose given. The total amount of pain medication administered per kg per day will be calculated by the study staff upon completion of the pain medication logs. Prior to surgery, a member of the study team will conduct a brief standard training session for parents to teach them how to correctly complete the medication log.
* Breakthrough pain: Patients who are randomized into the test intervention arm will receive ibuprofen (10mg/kg/day every 6-8 hours) after surgery. Patients who are randomized into the control intervention will receive hydrocodone-acetaminophen (0.15mg/kg/day every 4-6 hours). Both post-operative intervention groups in this study will have surgery for the same preoperative indications (adenotonsillitis or sleep disordered breathing). If patients experience pain that is not controlled with the specified intervention group medication, there will be a protocol in place for breakthrough pain, as indicated below. Surgeons will be blinded to the intervention arm. For patients who have pain that is not controlled by the randomized intervention, a breakthrough pain protocol will be enacted. The protocol is as follows:
* Test intervention arm

  1. Give hydrocodone-acetaminophen (0.15mg/kg/day hydrocodone) for pain score ≥6 no more than ever 6 hours. If uncontrolled pain, see next bullet point.
  2. Increase hydrocodone-acetaminophen dose to 0.2mg/kg/day hydrocodone per dose.
* Control intervention arm

  1. Increase dose of hydrocodone-acetaminophen to 0.2 mg/kg/day hydrocodone For pain score ≥ 6. If uncontrolled pain, see next bullet point.
  2. Ibuprofen 10mg/kg/day no more than every 6 hours. If uncontrolled pain, see next bullet point.
  3. Acetaminophen 10mg/kg/day every 6 hours as needed.

Implementation of the breakthrough pain protocol will be documented. In order to maintain surgeon blinding throughout the study, patient phone calls will be routed to the chief resident on call who will follow the above breakthrough pain protocol.

A study staff member, excluding the surgeon, will contact parents/caretakers on post-operative day 3 and post-operative day 7 to assist with medication log completion and answer medical questions.

ELIGIBILITY:
Inclusion Criteria:

* ≥4 and ≤17 years old
* Meeting criteria for tonsillectomy based on AAO-HNS clinical guidelines: Adenotonsillectomy is indicated for patients with recurrent adenotonsillitis and sleep disordered breathing. Both groups in this study will have surgery for the same preoperative indications

Exclusion Criteria:

* <4 or >17 years old
* Known bleeding diathesis (or family history of bleeding diathesis)
* Known allergy to any study medication
* participant/caregiver inability to understand or complete the required study documentation (pain scales, medication logs)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Rajan, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Randel A. AAO-HNS Guidelines for Tonsillectomy in Children and Adolescents. Am Fam Physician. 2011 Sep 1;84(5):566-73. No abstract available. PMID 21888309
- [Background] Marret E, Flahault A, Samama CM, Bonnet F. Effects of postoperative, nonsteroidal, antiinflammatory drugs on bleeding risk after tonsillectomy: meta-analysis of randomized, controlled trials. Anesthesiology. 2003 Jun;98(6):1497-502. doi: 10.1097/00000542-200306000-00030. No abstract available. PMID 12766664
- [Background] Lewis SR, Nicholson A, Cardwell ME, Siviter G, Smith AF. Nonsteroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database Syst Rev. 2013 Jul 18;2013(7):CD003591. doi: 10.1002/14651858.CD003591.pub3. PMID 23881651
- [Background] St Charles CS, Matt BH, Hamilton MM, Katz BP. A comparison of ibuprofen versus acetaminophen with codeine in the young tonsillectomy patient. Otolaryngol Head Neck Surg. 1997 Jul;117(1):76-82. doi: 10.1016/S0194-59989770211-0. PMID 9230328
- [Background] Mitchell RB, Kelly J. Behavior, neurocognition and quality-of-life in children with sleep-disordered breathing. Int J Pediatr Otorhinolaryngol. 2006 Mar;70(3):395-406. doi: 10.1016/j.ijporl.2005.10.020. PMID 16321451
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Hong SM, Cho JG, Chae SW, Lee HM, Woo JS. Coblation vs. Electrocautery Tonsillectomy: A Prospective Randomized Study Comparing Clinical Outcomes in Adolescents and Adults. Clin Exp Otorhinolaryngol. 2013 Jun;6(2):90-3. doi: 10.3342/ceo.2013.6.2.90. Epub 2013 Jun 14. PMID 23799166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between November 2014 and February 2016.
Pre-assignment Details: Eight of the 53 individuals who consented to taking part in the study did not meet eligibility criteria, resulting in 45 participants who began the intervention.
Groups:
- Ibuprofen: Participants randomized to receive ibuprofen (10mg/kg/day every 6-8 hours) after undergoing adenotonsillectomy.
- Hydrocodone-acetaminophen: Participants randomized to receive hydrocodone-acetaminophen (0.15mg/kg/day every 4-6 hours) after undergoing adenotonsillectomy.
Period: Overall Study
Arm/Group | Ibuprofen | Hydrocodone-acetaminophen
Started | 18 | 27
Completed | 9 | 8
Not Completed | 9 | 19
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 6 | 17

BASELINE CHARACTERISTICS:
Population: Children undergoing tonsillectomy who met all eligibility criteria and enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Hydrocodone-acetaminophen | Total
Number analyzed (Participants) | 18 | 27 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 27 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 17 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 27 | 45

OUTCOME MEASURES:

1. Primary Outcome: Faces Pain Score
Description: Using the Faces Pain Scale, the pediatric patient will indicate his/her pain level at scheduled intervals (7 times per day) for 14 days post-surgery.The Faces Pain Scale Revised is a dimensionless 10 point likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain. For this analysis, participant pain scores were summed and the mean per group was calculated. Total summed scores could range from 0 to 980.
Time Frame: 2 weeks after surgery
Population: Children who returned the completed the survey at two weeks post-surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen | Hydrocodone-acetaminophen
Number analyzed (Participants) | 10 | 8
units on a scale | 158.95 (9.33) | 219.94 (21.43)

2. Secondary Outcome: Number of Participants With Post-operative Bleeding
Description: The occurrence of post-operative bleeding at the surgical site for each participant will be assessed by review of the participant's study records and clinical records and by questioning the caregiver in follow-up. If postoperative bleeding has occurred, details of the episode of bleeding will also be obtained (requirement for surgical intervention, observation at home, or observation at the hospital).
Time Frame: 2 weeks after surgery
Population: All study participants are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen | Hydrocodone-acetaminophen
Number analyzed (Participants) | 18 | 27
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for two weeks following surgery.
Arm/Group | Ibuprofen | Hydrocodone-acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/27
Other Adverse Events (participants affected / at risk) | 1/18 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=18) | Hydrocodone-acetaminophen (N=27)
Hospitalization due to low oral intake and dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=18) | Hydrocodone-acetaminophen (N=27)
Emergency room visit due to bleeding (Surgical and medical procedures) | 1 (1) | 0 (0)
Emergency room visit due to pain (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Many participants did not completed the pain control survey, limiting the conclusions that can be made from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes